CLINICAL TRIAL: NCT01751984
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Efficacy and Safety of ETC-1002 in Subjects With Hypercholesterolemia and a History of Statin Intolerance
Brief Title: A Study of the Efficacy and Safety of ETC-1002 in Participants With Statin Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-006
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Hypercholesterolemia
Keywords: lipid-lowering drugs; statin intolerance
MeSH Terms: conditions — Hypercholesterolemia | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETC-1002 (Experimental): ETC-1002 treatment, once daily oral
  Interventions: Drug: ETC-1002
- Placebo (Placebo Comparator): Placebo treatment, once daily oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — Weeks 1-2, 60 milligrams per day (mg/day); Weeks 3-4, 120 mg/day; Weeks 5-6, 180 mg/day; Weeks 7-8, 240 mg/day
  Arms: ETC-1002
Drug: Placebo — Placebo once daily for 8 weeks
  Arms: Placebo

SUMMARY:
This study will assess the Low-Density Lipoprotein-Cholesterol (LDL-C) lowering efficacy and safety of ETC-1002 versus placebo in participants with hypercholesterolemia and a history of statin intolerance.

ELIGIBILITY:
Key Inclusion Criteria:

* A history of statin intolerance that began during statin treatment and resolved within 4 weeks of stopping the statin treatment
* For participants on current lipid-regulating drugs - LDL-C 100-220 milligrams per deciliter (mg/dL) and triglycerides <350 mg/dL (prior to wash-out of all lipid-regulating drugs and supplements)
* For participants not on current lipid-regulating drugs - LDL-C 115-270 mg/dL and fasting TG <400 mg/dL

Key Exclusion Criteria:

* Acute significant cardiovascular disease
* Poorly controlled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2012-10-04 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Esperion Therapeutics, Inc.
Locations (5):
- United States (5):
  - Hartford, Connecticut
  - Indianapolis, Indiana
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Knoxville, Tennessee

REFERENCES:
- [Result] Thompson PD, Rubino J, Janik MJ, MacDougall DE, McBride SJ, Margulies JR, Newton RS. Use of ETC-1002 to treat hypercholesterolemia in patients with statin intolerance. J Clin Lipidol. 2015 May-Jun;9(3):295-304. doi: 10.1016/j.jacl.2015.03.003. Epub 2015 Mar 19. PMID 26073387

RESULTS

PARTICIPANT FLOW:
Groups:
- ETC-1002: Participants initially received ETC-1002 60 milligrams (mg) once daily (QD) on Day 1 for 2 weeks, and then were titrated successively to 120 mg QD for 2 weeks, 180 mg QD for 2 weeks, and 240 mg QD for 2 weeks.
- Placebo: Participants received placebo QD on Day 1 for 8 weeks.
Period: Overall Study
Arm/Group | ETC-1002 | Placebo
Started | 37 | 19
Completed | 31 | 15
Not Completed | 6 | 4
Not completed — Adverse Event | 5 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Per Investigator/Sponsor/Regulatory Body | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Population, comprised of all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | ETC-1002 | Placebo | Total
Number analyzed (Participants) | 37 | 19 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] — Baseline was defined as the value from Week 0.
  years | 63.9 (5.42) | 60.4 (7.88) | 62.8 (6.51)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline was defined as the value from Week 0.
  Participants
    Female | 17 | 11 | 28
    Male | 20 | 8 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants] — Baseline was defined as the value from Week 0.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 2 | 0 | 2
    White | 35 | 19 | 54
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Calculated Low-density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] — Baseline was defined as the value from Week 0. Population: Only participants with available data were analyzed.
  milligrams per deciliter (mg/dL)
    number analyzed (Participants) | 36 | 19 | 55
    (all) | 175.7 (36.52) | 184.8 (32.53) | 178.9 (35.16)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 8 in Calculated Low-Density Lipoprotein-Cholesterol (LDL-C)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. Least square (LS) mean percent change from Baseline to Week 8 was based on an analysis of covariance (ANCOVA) model with effects of treatment and Baseline value as a covariate. Missing LDL-C values at Week 8 were imputed using the last observation carried forward (LOCF) procedure (only post-Baseline values were carried forward). A negative percent change from Baseline reflects clinical improvement.
Time Frame: Baseline; 8 weeks
Population: Modified Intent-to-Treat (mITT) Population: All randomized participants who received at least 1 dose of study medication and had a Baseline assessment and at least 1 post-Baseline assessment, excluding any assessments taken more than 2 days after a dose of study medication. The participant composition of this population could change depending on the parameter being analyzed. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 35 | 18
Percent Change | -32.0 (1.93) | -3.3 (2.69)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -28.7, 95% CI 2-sided [-35.4 to -22.1] — The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm

2. Secondary Outcome: Percent Change From Baseline to Weeks 2, 4, 6, and 8 in Calculated LDL-C
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline was based on an ANCOVA model with effects of treatment and Baseline value as a covariate. A negative percent change from Baseline reflects clinical improvement.
Time Frame: Baseline; Weeks 2, 4, 6, and 8
Population: Completers Population: All randomized participants who received at least 1 dose of study medication and had a Baseline assessment and an assessment at the specified time point, excluding any assessments taken more than 2 days after a dose of study medication. The participant composition of this population could change depending on the parameter being analyzed. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 36 | 18
Percent Change
  Week 2: number analyzed (Participants) | 34 | 18
  Week 2 | -19.5 (1.83) | -1.4 (2.52)
  Week 4: number analyzed (Participants) | 30 | 15
  Week 4 | -31.0 (1.50) | -1.0 (2.12)
  Week 6: number analyzed (Participants) | 31 | 15
  Week 6 | -32.6 (2.28) | -3.8 (3.28)
  Week 8: number analyzed (Participants) | 26 | 13
  Week 8 | -32.6 (2.48) | -4.0 (3.51)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -18.0, 95% CI 2-sided [-24.3 to -11.8] — Estimation from Week 2. The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm
Statistical Analysis 2: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -30.0, 95% CI 2-sided [-35.2 to -24.7] — Estimation from Week 4. The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm
Statistical Analysis 3: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -28.8, 95% CI 2-sided [-36.9 to -20.8] — Estimation from Week 6. The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm
Statistical Analysis 4: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -28.5, 95% CI 2-sided [-37.2 to -19.8] — Estimation from Week 8. The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm

3. Secondary Outcome: Percent Change From Baseline to Week 8 in High-Density Lipoprotein-Cholesterol (HDL-C)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline to Week 8 was based on an ANCOVA model with effects of treatment and Baseline value as a covariate. Missing values at Week 8 were imputed using the LOCF procedure (only post-Baseline values were carried forward). A negative percent change from Baseline reflects clinical improvement.
Time Frame: Baseline; 8 weeks
Population: mITT Population. The participant composition of this population could change depending on the parameter being analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 36 | 18
Percent Change | -8.2 (2.46) | -2.4 (3.51)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.1892, ANCOVA; Least squares mean difference = -5.8, 95% CI 2-sided [-14.5 to 2.9] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percent Change From Baseline to Week 8 in Non-HDL-C
Description: as for outcome 3
Time Frame: Baseline; 8 weeks
Population: mITT Population. The participant composition of this population could change depending on the parameter being analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 36 | 18
Percent Change | -25.4 (2.04) | -4.4 (2.88)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -20.9, 95% CI 2-sided [-28.0 to -13.9] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percent Change From Baseline to Week 8 in Total Cholesterol
Description: as for outcome 3
Time Frame: Baseline; 8 weeks
Population: mITT Population. The participant composition of this population could change depending on the parameter being analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 36 | 18
Percent Change | -22.2 (1.64) | -3.7 (2.32)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Least squares mean difference = -18.4, 95% CI 2-sided [-24.2 to -12.7] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Percent Change From Baseline to Week 8 in Triglycerides
Description: as for outcome 3
Time Frame: Baseline; 8 weeks
Population: mITT Population. The participant composition of this population could change depending on the parameter being analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 36 | 18
Percent Change | 11.2 (6.34) | -7.4 (8.98)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.0962, ANCOVA; Least squares mean difference = 18.7, 95% CI 2-sided [-3.5 to 40.8] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percent Change From Baseline to Week 8 in Apolipoprotein B
Description: as for outcome 3
Time Frame: Baseline; 8 weeks
Population: mITT Population. The participant composition of this population could change depending on the parameter being analyzed. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 29 | 14
Percent Change | -19.7 (2.61) | -4.4 (3.77)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.0019, ANCOVA; Least squares mean difference = -15.3, 95% CI 2-sided [-24.6 to -6.0] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percent Change From Baseline to Week 8 in Apolipoprotein AI
Description: as for outcome 3
Time Frame: Baseline; 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 29 | 14
Percent Change | -4.2 (2.04) | 0.1 (2.98)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.2555, ANCOVA; Least squares mean difference = -4.2, 95% CI 2-sided [-11.7 to 3.2] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percent Change From Baseline to Week 8 in Lipoprotein (a)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline to Week 8 was based on an ANCOVA model with effects of treatment and Baseline value as a covariate. Data are based on the participant's last post-Baseline value. Only those participants having a valid assessment at Baseline and each subsequent time point were included in the summaries at that time point. Lipoprotein (a) results indicated as <3 in the laboratory data were set to 3 for purposes of analysis. A negative percent change from Baseline reflects clinical improvement.
Time Frame: Baseline; 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 29 | 14
Percent Change | 10.4 (5.78) | -1.2 (8.32)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.2563, ANCOVA; Least squares mean difference = 11.7, 95% CI 2-sided [-8.8 to 32.1] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percent Change From Baseline to Week 8 in High-Sensitivity C-Reactive Protein (hsCRP)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline to Week 8 was based on an ANCOVA model with effects of treatment and Baseline value as a covariate. Data were based on the participant's last post-Baseline value. Only those participants having a valid assessment at Baseline and each subsequent time point were included in the summaries at that time point. hsCRP results indicated as <0.2 in the laboratory data were set to 0.2 for purposes of analysis. A negative percent change from Baseline reflects clinical improvement.
Time Frame: Baseline; 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 28 | 14
Percent Change | -22.6 (11.77) | 1.1 (16.74)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.2565, ANCOVA; Least squares mean difference = -23.7, 95% CI 2-sided [-65.4 to 18.0] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percent Change From Baseline to Week 8 in Free Fatty Acids (FFA)
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the value from Week 0. LS mean percent change from Baseline to Week 8 was based on an ANCOVA model with effects of treatment and Baseline value as a covariate. Data were based on the participant's last post-Baseline value.
Time Frame: Baseline; 8 weeks
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 28 | 14
Percent Change | 14.3 (7.99) | 10.4 (11.31)
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p = 0.7760, ANCOVA; Least squares mean difference = 4.0, 95% CI 2-sided [-24.1 to 32.0] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Number of Participants Achieving Their National Cholesterol Education Program Adult Treatment Panel III (NCEP ATPIII) LDL-C Goal (<100 Milligrams Per Deciliter [mg/dL]) After 8 Weeks of Treatment
Description: Participants were analyzed to evaluate the LDL-C target of <100 mg/dL for high risk participants with cardiovascular diseases. Missing values at Week 8 were imputed using the LOCF procedure (only post-Baseline values were carried forward).
Time Frame: Baseline; up to 8 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 34 | 17
Participants
  Week 8: Achieved LDL-C Goal | 21 | 0
  Week 8: Did Not Achieve LDL-C Goal | 13 | 17
Statistical Analysis 1: Comparison: ETC-1002 vs Placebo; Test type: Superiority; p < 0.0001, Fisher Exact — Based on Fisher's exact test comparing the proportion of participants who achieved LDL-C goal at Week 8 (End of Study) in the ETC-1002 and placebo groups; Clopper-Pearson methodology = 61.8, 95% CI 2-sided [45.4 to 78.1] — ETC-1002 minus placebo for the proportion of participants who achieved LDL-C goal at Week 8 (End of Study). The confidence interval was based on a normal approximation to the binomial distribution

13. Secondary Outcome: Number or Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) that began or worsened in severity after the first dose of study medication, occurring up to 30 days after the last dose of study medication.
Time Frame: up to 8 weeks
Population: Safety Population: all randomized participants who received at least 1 dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 37 | 19
Participants | 26 | 15

14. Secondary Outcome: Number of Participants With Muscle-Related TEAEs
Description: TEAEs were defined as AEs that began or worsened in severity after the first dose of study medication, occurring up to 30 days after the last dose of study medication.
Time Frame: up to 8 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 | Placebo
Number analyzed (Participants) | 37 | 19
Participants | 12 | 7

ADVERSE EVENTS:
Time Frame: up to 8 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began or worsened in severity after the first dose of study medication, occurring up to 30 days after the last dose of study medication, are reported. The analysis was performed using the Safety Population, comprised of all randomized participants who received at least 1 dose of study medication.
Arm/Group | ETC-1002 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/19
Other Adverse Events (participants affected / at risk) | 19/37 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 (N=37) | Placebo (N=19)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 (N=37) | Placebo (N=19)
Eye Swelling (Eye disorders) | 0 | 1
Change Of Bowel Habit (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 2 | 1
Oedema (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Rhinovirus Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 4
Urinary Tract Infection (Infections and infestations) | 3 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1
White Blood Cells Urine Positive (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5 | 1
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dizziness Postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No